CLINICAL TRIAL: NCT01362205
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Dexmedetomidine (Precedex®), With Lorazepam Rescue, for the Management of Severe Alcohol Withdrawal Syndrome (AWS) and Alcohol Withdrawal Delirium (AWD)
Brief Title: Dexmedetomidine (Precedex®) for Severe Alcohol Withdrawal Syndrome (AWS) and Alcohol Withdrawal Delirium (AWD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DSMB recommendation for slow enrollment
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Ivor Douglas, Professor of Medicine, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COMIRB 09-0822
Record Dates: First submitted 2010-05-24; First posted 2011-05-30 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Withdrawal Delirium; Alcohol Withdrawal Associated Autonomic Hyperactivity; Alcohol Withdrawal Hallucinosis; Alcohol Withdrawal-Induced Delirium Tremens
Keywords: Severe Alcohol Withdrawal Delirium Tremens
MeSH Terms: conditions — Alcohol Withdrawal Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine titrated to achieve predefined goals on selected components of the MINDS score using the minimum amount of medication possible. Blinded study medication will be started at a rate determined by the MINDS score. The maximum infusion rate is 1.4 μg/kg per hour. Uncontrolled SAWS/D symptoms, will be treated with open label lorazepam according to the MINDS score algorithm. Persistent SAWS/D symptoms despite maximum infusion rate of study medication treatment limiting symptoms while receiving higher infusion rates of study medication, ancillary therapies will be administered according to the MINDS score algorithm, at the discretion of the treating physician.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Blinded placebo study drug administration in equal volume per hour as active study medication arm.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Placebos — Inactive placebo (normal saline)
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled, parallel-group study of dexmedetomidine versus placebo, with lorazepam rescue, for the management of severe alcohol withdrawal syndrome (AWS) and alcohol withdrawal delirium (AWD) in critically ill adults.

The investigators hypothesize that the integration of dexmedetomidine (Precedex®) with usual therapy for the management of severe alcohol withdrawal syndrome (AWS) and alcohol withdrawal delirium/delirium tremens (AWD) in critically ill adult patients will reduce the time to resolution of AWS/AWD, increase the number of delirium-free and ventilator-free days in the first 28 days of hospitalization, reduce the length of ICU and hospital stays, and improve neurocognitive and quality of life scores on hospital discharge.

DETAILED DESCRIPTION:
Severe alcohol withdrawal syndrome (AWS) and alcohol withdrawal delirium (AWD) are frequent principal indication/s for admission to intensive care units. Additionally, unanticipated alcohol withdrawal complicates other critical illnesses and peri-operative states. Alcohol intoxication and withdrawal syndrome are characterized by classic symptoms of adrenergic activation, psychiatric agitation including seizures, as well as metabolic and respiratory dysfunction. The majority of patients with severe AWS are effectively managed with combinations of benzodiazepine (BZD) sedatives (e.g. lorazepam) and butyrophenone antipsychotics (e.g. haloperidol) and require intensive care admission for 2-3 days. However, almost 25% of patients with SAWS have a prolonged critical care course, often complicated by respiratory failure and associated with excessive sedation and risk for complications such as ventilator-associated pneumonia (VAP). AWS is frequently difficult to manage with usual care including benzodiazepines. Additionally, while intermittent bolus dose sedation is recommended for AWS, high dose BZD alone is associated with excessive respiratory suppression and metabolic acidosis. Such therapy increases the likelihood of respiratory failure with its attendant complications of hospital acquired pneumonia and sepsis. Further, patients with underlying chronic liver disease are at greater risk for prolonged sedative effects of BZD and progression of hepatic encephalopathy. The requirement for mechanical ventilation additionally prolongs the course of treatment for AWD because of the need for prolonged sedation. Strategies to control AWS/AWD that control symptoms but avoid adverse effects of excessive respiratory suppression are anticipated to improve the short and medium-term outcomes of AWS.

BZD infusions have also been shown by several investigators to result in excessive and prolonged sedation. However, reasonable alternatives for effective control of psychomotor and adrenergic activation have until recently, been unavailable. The centrally acting alpha-2 receptor agonist, clonidine has been suggested as a useful adjunctive therapy to BZD. However, clonidine is only a mild sedative and can result in significant hemodynamic compromise. By contrast, dexmedetomidine (Precedex), a more potent alpha-2 receptor agonist, is potentially a more effective adjunctive therapy. Precedex is currently marketed in the USA for short-term use as a potent peri-operative sedative and analgesic. This agent has a short circulating half-life and has significantly fewer hemodynamic side effects than clonidine. In addition to its cardiovascular properties, dexmedetomidine possesses anxiolytic, hypnotic/sedative, anesthetic-sparing and analgesic actions and is devoid of significant respiratory depressant effects.

Precedex has been shown to be a safe and effective single agent sedative for critically ill medical and surgical patients in prolonged infusions up to thirty days and is associated with significantly lower incidence of delirium than sedation with the benzodiazepine, midazolam. Preclinical experience and case reports suggest anecdotally Precedex may be of particular benefit in patients with SAWS.

Measures of sedation and delirium will be assessed with the Minnesota Detoxification Scale (MINDS) derived for use in critically ill adults from the validated Clinical Institute Withdrawal Assessment (CIWA-r) scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 years or older, with severe AWS or AWD per DSM-IV definitions (below) requiring admission to the ICU for medical management
* Ability to provide informed consent (via a proxy decision maker or patient).
* Within 96 hours of ICU admission.
* Meets DSM-IV diagnostic criteria for 291.8 Alcohol Withdrawal Syndrome:

  * Cessation of (or reduction in) alcohol use that has been heavy and prolonged.
  * Two (or more) of the following, developing within several hours to a few days after Criterion A:

    1. autonomic hyperactivity (e.g., sweating or pulse rate greater than 100)
    2. increased hand tremor
    3. insomnia
    4. nausea or vomiting
    5. transient visual, tactile, or auditory hallucinations or illusions
    6. psychomotor agitation
    7. anxiety
    8. grand mal seizures
* The symptoms are not due to a general medical condition and are not better accounted for by another mental disorder.

AND Meets DSM-IV diagnostic criteria for 291.0 Alcohol Intoxication or Withdrawal Delirium

* Disturbance of consciousness
* A change in cognition
* The disturbance develops over a short time and can fluctuate
* Onset is temporal associated with Alcohol Withdrawal Syndrome

Exclusion Criteria:

* Age < 18 years
* Physician anticipates ICU transfer orders in less than 12 hours from time of consent.
* Recent traumatic brain injury
* Active status epilepticus
* Pregnancy or lactation
* Known allergy or adverse response to any of the study medications
* Requiring glucocorticoid therapy for treatment of acute hepatitis or Stage III (advanced) decompensated liver failure and encephalopathy
* Trauma or burns as admitting diagnoses
* Neuromuscular blockade other than for intubation
* Epidural or spinal analgesia
* General anesthesia 24 hours prior to, or planned after, the start of study drug infusion
* Serious central nervous system pathology (acute stroke, uncontrolled seizures, severe dementia),
* Unstable angina or acute myocardial infarction
* Left ventricular ejection fraction less than 30%
* Heart rate less than 50/min
* Second- or third degree heart block
* Systolic blood pressure less than 90 mm Hg despite continuous infusions of 2 vasopressors before the start of study drug infusion.
* Previous randomization into this study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor S Douglas, MD, FRCP, Principal Investigator — Denver Health Medical Center
Locations (7):
- United States (7):
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Denver Health Medical Center, Medical ICU, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Anthony Hospital, Lakewood, Colorado
  - Louisiana State University, New Orleans, Louisiana
  - Ben Taub Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Darrouj J, Puri N, Prince E, Lomonaco A, Spevetz A, Gerber DR. Dexmedetomidine infusion as adjunctive therapy to benzodiazepines for acute alcohol withdrawal. Ann Pharmacother. 2008 Nov;42(11):1703-5. doi: 10.1345/aph.1K678. Epub 2008 Sep 9. PMID 18780809
- [Background] Rovasalo A, Tohmo H, Aantaa R, Kettunen E, Palojoki R. Dexmedetomidine as an adjuvant in the treatment of alcohol withdrawal delirium: a case report. Gen Hosp Psychiatry. 2006 Jul-Aug;28(4):362-3. doi: 10.1016/j.genhosppsych.2006.03.002. PMID 16814639
- [Background] Maccioli GA. Dexmedetomidine to facilitate drug withdrawal. Anesthesiology. 2003 Feb;98(2):575-7. doi: 10.1097/00000542-200302000-00041. No abstract available. PMID 12552220

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: Dexmedetomidine titrated to achieve predefined goals on selected components of the MINDS score using the minimum amount of medication possible. Blinded study medication will be started at a rate determined by the MINDS score. The maximum infusion rate is 1.4 μg/kg per hour. Uncontrolled SAWS/D symptoms, will be treated with open label lorazepam according to the MINDS score algorithm. Persistent SAWS/D symptoms despite maximum infusion rate of study medication treatment limiting symptoms while receiving higher infusion rates of study medication, ancillary therapies will be administered according to the MINDS score algorithm, at the discretion of the treating physician.
  Dexmedetomidine: See arm details
- Placebo: Blinded placebo study drug administration in equal volume per hour as active study medication arm.
  Placebo: Sterile, clear saline 0.9%
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 22 | 27
Completed | 22 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 22 | 27 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.54) | 48.2 (11.82) | 47.4 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 16 | 24 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 19 | 24 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: The Length of ICU Stay Defined as the Time Between Randomization and ICU Transfer Orders.
Time Frame: up to 28 days in hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
hours | 79.2 [43.9 to 134.6] | 104.9 [63.7 to 183.1]
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Test type: Other; p = 0.2454, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Average MINDS Score
Description: Minnesota Detoxification Scale (MINDS) min score 0, max score 46. The higher the score, the worse the symptoms of AWS/AWD.
Time Frame: up to 28 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
units on a scale | 8.2 [4.6 to 11.0] | 9.4 [7.8 to 11.6]

3. Secondary Outcome: The Number of CAM-ICU Negative Days After Randomization.
Description: The Confusion Assessment Method (CAM)-ICU is a validated instrument used to detect the presence or absence of delirium in the ICU. A delirium free day is counted for any day a patient is negative by the CAM-ICU. The higher the number of CAM-ICU negative days indicates the more days a patient was able to think clearly.
Time Frame: up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
days | 0.3 [0.0 to 0.5] | 0.3 [0.1 to 0.7]

4. Secondary Outcome: Number of Ventilator Free Days After Randomization.
Description: A ventilator day is counted for any use of invasive mechanical ventilation during a calendar day
Time Frame: up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
days | 27.5 [25.0 to 28.0] | 28.0 [26.0 to 28.0]

5. Secondary Outcome: The Length in Days of the Hospital Stay
Description: A hospital day is counted for any time on a calendar day the patient is admitted to the hospital. Hospital days are inclusive of ICU days.
Time Frame: up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
days | 8.0 [5.0 to 13.0] | 12.0 [6.0 to 16.0]

6. Secondary Outcome: Scores at Hospital Discharge on the Mini Mental Exam.
Description: The Mini Mental State Examination or Folstein test is a validated 30-point questionnaire used to measure cognitive impairment (min score 0, max score 30). A score of 24 points (out of a max of 30) indicates normal cognition, less than or equal to 9 points indicates severe impairment, 10-18 indicates moderate impairment and 19-23 mild impairment.
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
units on a scale | 25.8 (2.53) | 23.1 (6.09)

7. Secondary Outcome: Scores at Hospital Discharge on the Beck Depression Inventory.
Description: The Beck Depression Inventory is a validated questionnaire used to measure severity of depression (min score 0, max score 63). The higher the score the greater the severity of depression. A score of 30-63 indicates severe depression, 19-29 moderate depression, 10-18 mild depression and 0-9 minimal depression.
Time Frame: Up to 28 days.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
units on a scale | 26.5 (9.14) | 21.4 (10.95)

8. Secondary Outcome: Scores at Hospital Discharge on the Beck Anxiety Inventory
Description: The Beck Anxiety Inventory is a validated questionnaire used to measure severity of anxiety (min score 0, max score 63). The higher the score the greater the severity of anxiety. A score of 30-63 indicates severe anxiety, 17-29 moderate anxiety, 10-16 mild anxiety and 0-9 minimal anxiety.
Time Frame: Up to 28 days.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
units on a scale | 30.3 (10.83) | 21.6 (11.55)

9. Secondary Outcome: Scores at Hospital Discharge on the PTSD Civilian Checklist
Description: PTSD checklist consists of 17 questions graded on a scale of 1 to 5. The PTSD score is comprised from the sum of the scores 17 questions. The PTSD score has possible values from to 17 to 85 with higher values indicating greater symptom severity.
Time Frame: Up to 28 days
Population: The number of participants analyzed was lower than the total included as many patients were discharged quickly upon resolution of altered mental status when a research team member was unavailable to administer the questionnaires.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 8 | 12
units on a scale | 45.5 [39.0 to 59.5] | 32.5 [27.5 to 37.0]

10. Secondary Outcome: Resource Utilization Costs Associated With This Hospitalization Billed by Physicians.
Time Frame: up to 28 Days
Measure: Median (Inter-Quartile Range); unit: Dollar (United States)
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 27
Dollar (United States) | 3482 [2068 to 9326] | 4461 [2926 to 8001]

11. Secondary Outcome: Resource Utilization Costs Associated With This Hospitalization Billed by Facility.
Time Frame: Up to 28 days
Population: The overall number of participants analyzed is less than the number randomized as data was not available for research use at many of the participating institutions.
Measure: Median (Inter-Quartile Range); unit: USD
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 17 | 23
USD | 81234 [51437 to 137272] | 91651 [67341 to 132458]

ADVERSE EVENTS:
Time Frame: The first 28 days of hospitalization after randomization.
Description: One subject randomized to the dexmedetomidine group did not receive study drug and so was excluded from the adverse event analysis. The total number of subjects included in the adverse event analysis in the dexmedetomidine decreased from 22 to 21.
Arm/Group | Dexmedetomidine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/27
Serious Adverse Events (participants affected / at risk) | 5/21 | 3/27
Other Adverse Events (participants affected / at risk) | 12/21 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine (N=21) | Placebo (N=27)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Osmotic demyelination syndrome (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine (N=21) | Placebo (N=27)
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 4
Bradycardia (Cardiac disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Oedema peripheral (General disorders) | 6 | 11
Pyrexia (General disorders) | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 3
Haemoglobin decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 1 | 3
Protein total decreased (Investigations) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 5 | 13
Hypotension (Vascular disorders) | 6 | 4

LIMITATIONS AND CAVEATS:
Early termination due to slow enrollment leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No